CLINICAL TRIAL: NCT04317014
Title: Polymorphisms in Obesity-related Genes Are Associated With Risk of Early Puberty in Han Chinese Girls
Brief Title: the Association Between Obesity and Early Puberty
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Di Li, post doctor, Shenzhen Center for Disease Control and Prevention
Other Study IDs: szCDC_2
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Early Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: early puberty girls of Han Chinese
- controls: normal development girls of Han Chinese

SUMMARY:
childhood obesity and early puberty are closely related, but existing reports usually focus on their relationship from the perspective of phenotype. This study was designed to investigate the association between obesity-related genic polymorphisms and the risk of early puberty in Chinese Han girls.

DETAILED DESCRIPTION:
the genotypes of obesity-related SNPs were determined and the unstimulated luteinizing hormone, follicle stimulating hormone and estradiol levels were also detected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of central precocious puberty or early and fast puberty.

Exclusion Criteria:

* The participants who were not the first visit to the hospital and had been treated before.
* The participants who were with endocrine disorders.

Ages: 7 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Chinese Han girls from Shenzhen Children's Hospital or monitoring schools in Shenzhen
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
genotypes of SNPs in the obesity-related genes | 3 months
  the obesity-related SNPs in the LRRN6C, MAF, CYP27A1 and ETV5 genes are selected and the genotypes of these SNPs are determined with a MassARRAY system.